CLINICAL TRIAL: NCT04721353
Title: Pilot Study to Assess the Feasibility of Prazosin for Cannabis Use Disorder in Individuals With or Without Post-traumatic Stress Disorder
Brief Title: Reducing Cannabis Overuse With Prazosin
Acronym: ReCOUP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: University of Washington (Other); VA Mental Illness Research, Education and Clinical Centers (U.S. Federal Agency)
Responsible Party: Principal Investigator, Garth Terry, Assistant Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010457
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cannabis Dependence; Posttraumatic Stress Disorder; Cannabis Use Disorder
Keywords: Prazosin; Cannabis
MeSH Terms: conditions — Marijuana Abuse; Stress Disorders, Post-Traumatic | interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: Open-label study of prazosin for treatment of cannabis use disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-label prazosin treatment (Experimental): Open-label administration of prazosin
  Interventions: Drug: Prazosin Hydrochloride

INTERVENTIONS:
Drug: Prazosin Hydrochloride — prazosin hydrochloride oral 1-25 mg/day
  Other Names: minipress

SUMMARY:
Cannabis use disorder (CUD) is a significant and expanding health problem, and no FDA approved treatments are currently available. Persons with posttraumatic stress disorder (PTSD) may use cannabis to help control symptoms. Relief from PTSD insomnia, nightmares, anxiety, and preoccupying thoughts have been reported as troublesome symptoms targeted by cannabis users. Risks from cannabis use by individuals with PTSD have been reported. Chronic use of cannabis can lead to tolerance, requiring increased use for symptom relief, and withdrawal symptoms upon stopping. CUD is more frequent and severe in those with PTSD than those without. Many symptoms of cannabis withdrawal overlap with troubling symptoms of PTSD and thus may be interpreted as a relapse of PTSD symptoms. Those attempting to reduce or stop cannabis use may experience cannabis withdrawal symptoms including insomnia and distressing dreams, anxiety, irritability, and/or excessive sweating that they may misattribute to re-emerging or untreated PTSD symptoms.

Excessive brain adrenaline activity is arguably the best-described neurobiological contribution to the pathophysiology of PTSD. Prazosin, a drug that blocks the negative effects of brain adrenaline, has demonstrated effectiveness in robustly reducing PTSD-related nightmares and sleep disturbance in active duty Servicemembers and recently discharged combat Veterans in most, but not all, clinical trials, as well as in civilians with non-combat trauma. Clinically, the investigators have observed that several patients with PTSD using cannabis to treat insomnia and/or trauma-related nightmares and wanting to reduce their cannabis use were able to achieve reduction or cessation of cannabis use once they were treated with an effective dose of prazosin. Therefore, we have wondered if prazosin may provide sufficient treatment of PTSD symptoms otherwise targeted by cannabis, supporting those individuals' efforts to reduce cannabis use.

This open-label pilot study aims to study the feasibility of prazosin as a treatment for CUD in individuals with or without comorbid PTSD, and to evaluate if additional research on a larger scale is warranted.

DETAILED DESCRIPTION:
This pilot study aims to assess the feasibility of prazosin as a treatment for CUD in individuals with or without comorbid PTSD, and to evaluate if additional research on a larger scale is warranted. In particular, the investigators will evaluate their ability to recruit and retain individuals with CUD, evaluate their ability to quantify cannabis use and associated clinical outcomes, and objectively measure cannabis use in context of a clinical trial.

Although the investigators have ample experience recruiting Veterans and non-Veterans with and without PTSD for prazosin clinical trials of similar duration, they have never recruited treatment-seeking CUD participants. Treatment studies in cannabis users are known to have approximately 30% drop out rate, and thus gaining experience in recruitment and retention is critical prior to investment in larger studies.

Specific Aim 1: Assess the feasibility of recruitment and retention of participants for a clinical trial using prazosin as a treatment of CUD.

The investigators will recruit 20 treatment seeking individuals with CUD (10 with and 10 without PTSD) for 12-week open label treatment of prazosin. Given their experience conducting studies in Veterans and non-Veterans with and without PTSD and/or alcohol use disorder (AUD) achieving 61-83% retention at end of treatment, the investigators anticipate that prazosin will be well tolerated in the study population. Participants will be asked to provide qualitative assessments of treatment acceptability, or reasons for early termination for those who drop out of the study before end of treatment, so that these issues can be addressed in future study design.

Specific Aim 2: Assess the feasibility of quantifying cannabis consumption by subjective self-report and objective urine and blood testing.

Quantification of cannabis use is complex and not standard within the field. Due to the multiple routes of cannabis self-administration, variable cannabinoid concentration in cannabis products, and variable tolerance and pharmacokinetics across cannabis users, the investigators seek to gain experience in quantifying cannabis use by self-report and objective testing, as these measures will directly affect their outcome assessments expected in a subsequent clinical trial design. The investigators will assess amount and frequency of cannabis used by self-report (i.e., typical grams consumed per day, number of sessions per day of use), tracked with regular semi-quantitative urine tests and validated by quantitative blood and urine testing at selected time points. Self-reported cannabis use will be assessed by the Quantification of Cannabis Consumption (QCC), a brief questionnaire designed and preliminarily tested by the investigators, and the timeline follow back (TLFB). Symptoms of CUD and cannabis withdrawal will be assessed with validated self-report measures. Semi-quantitative urine tests will provide a relatively inexpensive and rapid means of testing cannabis use. These measures will be compared against less frequent and fully quantitative urine and blood analysis using liquid chromatography-mass spectrometry (LC/MS). If self-report and semi-quantitative urine tests are consistent with those from LC/MS, then they will be utilized in subsequent clinical trials.

Exploratory Aims: The investigators will explore if prazosin administration is well tolerated and is associated with a reduction of cannabis withdrawal symptom severity and/or cannabis use. As there are no effective treatments for CUD, a reduction of cannabis use by at least 20% from baseline to end of treatment will be considered meaningful enough to warrant future study. In comparison, rates for attaining negative urine tests in two recent medication trials paired with contingency management or psychotherapy were 22% and 29%, respectively (with identical rates in placebo and treatment groups). Adverse events will be monitored and compared their frequencies to that experienced in prior studies of prazosin conducted by the investigators as an exploratory outcome. Additional exploratory outcomes include the comparison of cannabis use throughout the study between those with and without PTSD, and the reduction of PTSD-related nightmares in the PTSD group.

ELIGIBILITY:
Inclusion Criteria for all participants:

1. Men, women, and persons of all races and ethnic backgrounds are eligible.
2. Age 18 to 80 years inclusive
3. Ability to complete self-assessments and other clinical assessments in English
4. Meet criteria for CUD within the last 30 days
5. Report a minimum of 4 days a week or more of cannabis use (as assessed by 30 day TLFB at screening visit)
6. Have a positive cannabinoid urine test
7. Be in good general health
8. Persons of childbearing potential must agree to use an effective means of birth control.

   Inclusion Criteria for participants with CUD and PTSD:
9. Have a confirmed diagnosis on the Mini-International Neuropsychiatric Interview (MINI).

Exclusion Criteria for all participants:

1. Presence of a cognitive disorder
2. History of moderate or severe traumatic brain injury (mild traumatic brain injury is not exclusionary)
3. Current or past 3 months substance use disorder of any substance other than cannabis or tobacco (e.g., AUD, opioid use disorder)
4. Current and/or ongoing use of any substance other than cannabis, tobacco, or alcohol within the last 30 days
5. Current and/or ongoing use of synthetic cannabinoids (e.g., Spice, K2) within the last 30 days
6. Positive urine drug screen for any drug of abuse other than cannabis at screening visit
7. Persons of childbearing potential who are pregnant, planning to become pregnant, or nursing during the study period
8. Allergy or previous adverse reaction to prazosin or other alpha-1 adrenoceptor antagonist
9. Previously diagnosed but untreated severe sleep apnea
10. Psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal
11. Any unstable medical illness that may place the participant at increased risk in the judgment of the clinician
12. Potential participants who have been taking trazodone will undergo a 2-week washout period before beginning study treatment to reduce risk of priapism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | Approximately 2 weeks
  Proportion of potential participants referred to the study meeting inclusion/exclusion criteria and complete the baseline visit
Retention | 12 weeks
  Mean and median weeks participants remained in the study between baseline and end of treatment at week 12
Acceptability of participation | 16 weeks
  Total score from a 7-item exit questionnaire each with 5 point scale responses assessing: likelihood of repeat participation, difficulty of participation, difficulty of attending study visits, difficulty of taking study medication, satisfaction with study team, likelihood of referral, overall satisfaction of participation
Quantifying cannabis consumption | 16 weeks
  Regression comparison of semi-quantitative urine tetrahydrocannabinol (THC) metabolite and self-reported cannabis use by timeline follow back over the course of the study

SECONDARY OUTCOMES:
Treatment outcome (exploratory) | 16 weeks
  Change in cannabis consumption pre/post prazosin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Garth E Terry, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- See also: Study group website — https://www.mirecc.va.gov/visn20/research/ptsd-tbi-research.asp